CLINICAL TRIAL: NCT01085916
Title: Prevalence of Asthma and Rhinitis Symptoms Among Secondary School Students in Saudi Arabia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: King Abdulaziz Medical City (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dr Mohamed Ouda Al Anaezi, King Abdul Aziz Medical City, Riyadh, Saudi Arabia.
Other Study IDs: KingAbdulazizMC 001
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-02

CONDITIONS: Asthma; Rhinitis
Keywords: prevalence of asthma and Rhinitis symptoms among secondary school students in Saudi Arabia
MeSH Terms: conditions — Asthma; Rhinitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this cross-sectional survey study is to describe the prevalence of asthma and Rhinitis symptoms among secondary school students in Saudi Arabia.

DETAILED DESCRIPTION:
Cross sectional survey based on ISAAC protocol to characterize the symptoms of asthma and rhinitis and measure their frequency and its prevalence among secondary schools students (age 15 to 18 years, boys and girls) in Riyadh city, Saudi Arabia in period from 1st of April 2010 to 31st of May 2010.

The ISAAC protocol stated that the study population should consist of at least 3,000 students aged 15-18 years- in this case, enrolled in at least 40 randomly selected schools.

The 15-18 year age group was chosen because it is the age most adolescents go to school regularly, making data collection easier. Once requested by the research team, the education authority will provide a list of all secondary schools in Riyadh city and the number of students by school and their grades.

There are 400 secondary schools for boys and 400 school for girls (total number of boys and girls students 50,000).

A two stage stratified random sample of 4000 students will be selected out of secondary schools for boys and girls , Their ages range from 16 to 18 years.

ELIGIBILITY:
Inclusion Criteria:

* 15:18 year age group

Exclusion Criteria:

* Younger than 15 years or older than 18 years

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 4000 students will be selected out of secondary schools for boys and girls , Their ages range from 16 to 18 years.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-05 (Estimated)